CLINICAL TRIAL: NCT05013268
Title: The Efficacy and Safety of Tislelizumab Combined With Taxanes and Platinum as Neoadjuvant Therapy for Patients With Local Advanced Cervical Carcinoma， an Open Lable，Single-center, Exploratory Clinical Trial
Brief Title: Tislelizumab Plus TP as Neoadjuvant Therapy for Local Advanced Cervical Carcinoma
Acronym: TiTanec
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yan Shi, Associate professor, Ruijin Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TiTanec
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cervical Squamous Cell Carcinoma
MeSH Terms: interventions — tislelizumab; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus TP regimen as neoadjuvant therapy for local advanced cervical carcinoma (Experimental): Experimental:
  Tislelizumab, paclitaxel/docetaxel, cisplatin/carboplatin The subjects enrolled in this trial will receive tislelizumab 200mg ivgtt d1, paclitaxel (175mg/m2 ivgtt d1) or docetaxel (75mg/m2 ivgtt d1), cisplatin (75mg/m2 ivgtt d1) or carboplatin (AUC=5 ivgtt d1). The regimen will be repeated every 3 weeks for 3 cycles. Chemotherapy regimen will be selected by investigators.
  Subjects will be enrolled serially.
  Interventions: Drug: Tislelizumab, paclitaxel/docetaxel, cisplatin/carboplatin

INTERVENTIONS:
Drug: Tislelizumab, paclitaxel/docetaxel, cisplatin/carboplatin — * Drug: Tislelizumab 200mg, d1, ivgtt, every 3 weeks, for 3 cycles
  * Drug: Paclitaxel; docetaxel Dose: 175mg/m2 d1; 75mg/m2 d1, every 3 weeks, for 3 cycles Other Name: none
  * Drug: Cisplatin; Carboplatin Dose: 75mg/m2 d1; AUC=5, d1, every 3 weeks, for 3 cycles Other Name: none

SUMMARY:
The goal of this clinical trail is to investigate the efficacy and safety of PD-1 antibody Tislelizumab plus TP regimen (taxane combined with platinum) as neoadjuvant therapy for patients diagnosed as local advanced cervical carcinoma (FIGO staging IB2-IIB).

DETAILED DESCRIPTION:
This phase I study is being conducted to establish efficacy and safety of Tislelizumab plus TP regimen (taxane combined with platinum) as neoadjuvant therapy for patients diagnosed as local advanced cervical carcinoma (FIGO staging IB2-IIB).

All enrolled patients will receive same intervention. Treatment naïve patients who are diagnosed as local advanced cervical squamous cell carcinoma will receive Tislelizumab plus TP regimen before surgery for 3 cycles. After treatment, radiographic evaluation will be performed to assess clinical efficacy. Patients who have objective response will undergo radical surgery. Patients who are disease stable or progression will undergo radical chemoradiotherapy. The primary endpoint is major pathological response rate (MPR).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed cervical squamous cell carcinoma.
2. Clinical staging FIGO IB2-IIB, treatment naive.
3. Female patients aged≥18 years.
4. ECOG performance status 0 or 1, expected lifetime≥3 months.
5. Adequate organ function: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥90g/L, ALT/AST ≤2.5x ULN, Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
6. HBV infected patients (inactive/asymptomatic carrier, chronic or active) with HBV DNA<500IU/ml (or 2500 copies/ml).
7. Pregnancy test of female patients with fertile activity should be negative within 7 days before enrollment. Patients should keep contraception during treatment.
8. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. Pregnancy or children bearing potential.
2. brain or meningeal metastasis.
3. With second primary malignant diseases.
4. With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
5. With uncontrollable complications
6. Inadequate organ function
7. Known hypersensitivity reaction to any of the study drugs or components.

9. Other unsuitable conditions determined by investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  Major pathological response rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
Objective response rate (ORR) | Up to 30 days after last completion of neoadjuvant treatment
  Objective Response Rate is defined as the percentage of patients with a documented complete response or partial response (CR + PR) based on RECIST v1.1.
Relapse free survival (RFS) | Up to approximately 36 months
  Relapse free survival is defined as the time from surgery to first local, regional, or distant tumor recurrence or metastasis, or deaths.
Disease free survival (DFS) | Up to approximately 36 months
  disease-free survival (DFS) is defined as surgery until documented disease recurrence or death from any cause in all patients (ITT population) who undergo surgery
Adverse Events | Up to approximately 12 months
  All patients who have received at least one dose of treatment will be included in the safety analysis. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Overall survival (OS) | Up to approximately 60 months
  Overall survival is defined as the time from signing ICF until death from any cause.

OTHER OUTCOMES:
Biomarkers analysis | Up to approximately 12 months
  The association between biomarkers expression (eg. PD-L1 CPS) in primary tumor and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Shi, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No